CLINICAL TRIAL: NCT00306163
Title: Nebulizer Trial: Evaluation of the Influence of Particle Size of Aerosolized AMP on Bronchial Responsiveness in Patients With Asthma and the Effects of Treatment With Ciclesonide Versus Fluticasone.
Brief Title: Responsiveness of Lower Airways in Adult Patients (18-60 Years) With Stable Asthma After Treatment With Ciclesonide and Fluticasone Propionate (BY9010/NL-101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/NL-101
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Results first posted 2010-04-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; AMP; Ciclesonide; Fluticasone propionate
MeSH Terms: conditions — Asthma | interventions — ciclesonide; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ciclesonide 160 µg
  Interventions: Drug: Ciclesonide
- 2 (Active Comparator): Fluticasone 100 µg
  Interventions: Drug: Fluticasone

INTERVENTIONS:
Drug: Ciclesonide — inhaled Ciclesonide 160 µg, once daily in the morning
  Arms: 1
Drug: Fluticasone — inhaled Fluticasone 100 µg, twice daily
  Arms: 2

SUMMARY:
The aim of this study is to compare the responsiveness of lower airways in adult patients with stable asthma after treatment with ciclesonide and fluticasone propionate. Treatment medication will be administered as follows: ciclesonide will be inhaled once daily at one dose level, fluticasone propionate will be inhaled twice daily at one dose level. The study duration consists of a baseline period (5 weeks) and a treatment period (5 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* History of bronchial asthma
* FEV1 > 1.20 L
* Positive Skin Prick Test
* Not more than 500 mcg/day fluticasone propionate or equivalent for at least 28 days prior to baseline visit

Main Exclusion Criteria:

* Clinically relevant abnormal laboratory values
* Concomitant severe diseases, diseases expected to interfere with the outcome of the study and diseases which are contra-indications for the use of inhaled steroids
* Chronic obstructive pulmonary disease (COPD) and /or other relevant lung diseases
* One asthma exacerbation within 2 months or more than 3 exacerbations within the last year prior to baseline visit
* Current smokers or ex-smokers with more than 10 pack years, or having smoked within 1 year prior to baseline visit
* Positive response to saline challenge at baseline visits
* Positive bronchial hyperresponsiveness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana Pharma/Nycomed, RB Groningen, Netherlands

REFERENCES:
- [Derived] Cohen J, Postma DS, Douma WR, Vonk JM, De Boer AH, ten Hacken NH. Particle size matters: diagnostics and treatment of small airways involvement in asthma. Eur Respir J. 2011 Mar;37(3):532-40. doi: 10.1183/09031936.00204109. Epub 2010 Jul 1. PMID 20595155

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 101 subjects gave Informed Consent. 64 subjects did not enter or discontinued the study due to various reasons.
Groups:
- Ciclesonide: 160 µg, once daily
- Fluticasone: 100 µg, twice daily
Period: Overall Study
Arm/Group | Ciclesonide | Fluticasone
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide | Fluticasone | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Statistics for the total value were not available. The cited numbers are the results of manual calculations.
  years | 39.61 (10.50) [32.54 to 46.64] | 46.02 (9.80) [37.85 to 55.52] | 42.25 (10.16) [37.58 to 51.75]
Gender [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: PC20 AMP (Post-treatment Compared to Baseline)
Description: Mean change of Provocative concentration of Adenosine-5'-monophosphate (PC20 AMP) leading to a 20 percent decrease in Forced expiratory volume in one second (FEV1) between post-treatment and baseline using two different particle sizes. - Small particles = Mass mean aerodynamic diameter (MMAD) of approximately 1.04-1.08 micron - Large particles = MMAD of approximately 9.9-10.6 micron
Time Frame: Baseline and 5 weeks
Population: The analyses on treatment effects were performed on all subjects who reached a PC20<640mg/mL.
Measure: Mean (Standard Deviation); unit: Logarithm (mg/mL)
Arm/Group | Ciclesonide | Fluticasone
Number analyzed (Participants) | 11 | 12
Logarithm (mg/mL)
  Baseline PC20 small-particle AMP | 4.9 (3.7) | 5.2 (2.1)
  Baseline PC20 large-particle AMP | 3.7 (2.6) | 3.0 (2.4)
  Post-Treatment PC20 small-particle AMP | 6.6 (2.0) | 6.0 (2.7)
  Post-Treatment PC20 large-particle AMP | 4.5 (2.3) | 4.3 (2.4)

2. Secondary Outcome: Δ (FVC/SVC) at PC20 (AMP)
Description: Change between baseline and post-treatment of the ratio of Forced Vital Capacity (FVC) and Slow Vital Capacity at PC20. Measured with either small or large partical size AMP.
Time Frame: Baseline and 5 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Tolerability
Time Frame: 5 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ciclesonide | Fluticasone
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 2/19 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide (N=19) | Fluticasone (N=18)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Common cold (Infections and infestations) | 1 (1) | 0 (0)
Pain armpit (General disorders) | 0 (0) | 1 (1)
Inflammation of the throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days